CLINICAL TRIAL: NCT02752074
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled Study of Pembrolizumab (MK-3475) in Combination With Epacadostat or Placebo in Subjects With Unresectable or Metastatic Melanoma (Keynote-252 / ECHO-301)
Brief Title: A Phase 3 Study of Pembrolizumab + Epacadostat or Placebo in Subjects With Unresectable or Metastatic Melanoma (Keynote-252 / ECHO-301)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INCB 24360-301 (ECHO-301); 2015-004991-31 (EudraCT Number)
Record Dates: First submitted 2016-04-22; First posted 2016-04-26 (Estimated); Results first posted 2019-05-15 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Melanoma
Keywords: Melanoma; Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab; epacadostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pembrolizumab + Epacadostat (Experimental): Pembrolizumab + Epacadostat
  Interventions: Drug: pembrolizumab + epacadostat
- Pembrolizumab + Placebo (Active Comparator): Pembrolizumab + Placebo
  Interventions: Drug: pembrolizumab + placebo

INTERVENTIONS:
Drug: pembrolizumab + epacadostat — * Pembrolizumab will be administered intravenously every 3 weeks starting at Day 1 (Week 1)
  * Epacadostat will be administered orally daily starting at Day 1 (Week 1)
  Arms: Pembrolizumab + Epacadostat
Drug: pembrolizumab + placebo — * Pembrolizumab will be administered intravenously every 3 weeks starting at Day 1 (Week 1)
  * Placebo will be administered orally daily starting at Day 1 (Week 1)
  Arms: Pembrolizumab + Placebo

SUMMARY:
The purpose of the study is to assess the efficacy, safety, and tolerability when combining pembrolizumab with epacadostat or placebo in participants with unresectable or metastatic melanoma

ELIGIBILITY:
Inclusion Criteria:

* Have histologically or cytologically confirmed melanoma
* Have unresectable Stage III or Stage IV melanoma, as per AJCC staging system not amenable to local therapy
* A minimum of 1 measurable lesion by CT or MRI
* Provide a baseline tumor biopsy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1

Exclusion Criteria:

* Has received prior systemic treatment for unresectable or metastatic melanoma (except BRAF directed therapy)
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or IDO1 inhibitor or any other antibody or drug specifically targeting checkpoint pathways other than anti-CTLA-4 which is permitted in the adjuvant setting
* Has received prior adjuvant therapy, monoclonal antibody or an investigational agent or device within 4 weeks or 5 half-lives (whichever is longer)
* Has an active infection requiring systemic therapy
* Has known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known history of or is positive for Hepatitis B or Hepatitis C
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 706 (Actual)
Dates: Start 2016-06-21 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2019-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Jones, MD, Study Director — Incyte Corporation
Locations (129):
- United States (34):
  - Birmingham, Alabama
  - Scottsdale, Arizona
  - Little Rock, Arkansas
  - Los Angeles, California
  - San Francisco, California
  - Santa Barbara, California
  - Santa Monica, California
  - Aurora, Colorado
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Fort Lauderdale, Florida
  - Jacksonville, Florida
  - Ocala, Florida
  - West Palm Beach, Florida
  - Chicago, Illinois
  - Peoria, Illinois
  - Iowa City, Iowa
  - Kansas City, Kansas
  - Lutherville, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Fridley, Minnesota
  - Billings, Montana
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Rochester, New York
  - Charlotte, North Carolina
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Salt Lake City, Utah
  - Fairfax, Virginia
  - Spokane, Washington
- Australia (7):
  - Camperdown, New South Wales
  - Westmead, New South Wales
  - Wollstonecraft, New South Wales
  - Cairns, Queensland
  - Greenslopes, Queensland
  - Kurralta Park, South Australia
  - Melbourne, Victoria
- Belgium (2):
  - Brussels
  - Ghent
- Canada (4):
  - North Vancouver, British Columbia
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Chile (2):
  - Santiago
  - Viña del Mar
- Denmark (3):
  - Aarhus
  - Herlev
  - Odense C
- France (9):
  - Bordeaux
  - Lille
  - Marseille
  - Paris
  - Pierre-Bénite
  - Reims
  - Rennes
  - Toulouse
  - Villejuif
- Germany (5):
  - Buxtehude
  - Essen
  - Hanover
  - Kiel
  - Tübingen
- Ireland (3):
  - Cork
  - Dublin
  - Galway
- Ramat Gan, Israel
- Italy (6):
  - Bergamo
  - Genova
  - Milan
  - Napoli
  - Padua
  - Siena
- Japan (17):
  - Susono, Sunto-gun
  - Asahikawa
  - Chūō
  - Fukuoka
  - Kagoshima
  - Kumamoto
  - Kurume
  - Kyoto
  - Matsumoto
  - Nagoya
  - Niigata
  - Okayama
  - Osaka
  - Sapporo
  - Sendai
  - Tokyo
  - Tsukuba
- Mexico (4):
  - Chihuahua City
  - Distrito Federal
  - Mexico City
  - Monterrey
- Netherlands (2):
  - Amsterdam
  - Nijmegen
- New Zealand (2):
  - Dunedin
  - Tauranga
- Warsaw, Poland
- Russia (3):
  - Istra
  - Moscow
  - Saint Petersburg
- South Africa (5):
  - Johannesburg, Gauteng
  - Sandton, Gauteng
  - Groenkloof, Pretoria
  - Cape Town, Western Cape
  - Kraaifontein
- Seoul, South Korea
- Spain (8):
  - Donostia / San Sebastian, Guipuzcoa
  - A Coruña
  - Barcelona
  - Donostia / San Sebastian
  - Madrid
  - Pamplona
  - Seville
  - Valencia
- Sweden (4):
  - Gothenburg
  - Lund
  - Stockholm
  - Uppsala
- Switzerland (3):
  - Zurich, Canton of Zurich
  - Geneva
  - Lausanne
- United Kingdom (3):
  - Edinburgh
  - London
  - Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Long GV, Dummer R, Hamid O, Gajewski TF, Caglevic C, Dalle S, Arance A, Carlino MS, Grob JJ, Kim TM, Demidov L, Robert C, Larkin J, Anderson JR, Maleski J, Jones M, Diede SJ, Mitchell TC. Epacadostat plus pembrolizumab versus placebo plus pembrolizumab in patients with unresectable or metastatic melanoma (ECHO-301/KEYNOTE-252): a phase 3, randomised, double-blind study. Lancet Oncol. 2019 Aug;20(8):1083-1097. doi: 10.1016/S1470-2045(19)30274-8. Epub 2019 Jun 17. PMID 31221619

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 135 centers in 23 countries
Groups:
- Pembrolizumab + Epacadostat: Pembrolizumab will be administered intravenously every 3 weeks starting at Day 1 (Week 1). Epacadostat will be administered orally daily starting at Day 1 (Week 1).
- Pembrolizumab + Placebo: Pembrolizumab will be administered intravenously every 3 weeks starting at Day 1 (Week 1). Placebo will be administered orally daily starting at Day 1 (Week 1).
Period: Overall Study
Arm/Group | Pembrolizumab + Epacadostat | Pembrolizumab + Placebo
Started | 354 | 352
Treated | 353 | 352
Completed | 198 | 209
Not Completed | 156 | 143
Not completed — Lost to Follow-up | 1 | 4
Not completed — Death | 146 | 129
Not completed — Withdrawal by Subject | 9 | 10

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) population: consists of all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + Epacadostat | Pembrolizumab + Placebo | Total
Number analyzed (Participants) | 354 | 352 | 706
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 183 | 193 | 376
  ≥ 65 years | 171 | 159 | 330
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137 | 146 | 283
  Male | 217 | 206 | 423
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 27 | 63
  Not Hispanic or Latino | 302 | 306 | 608
  Unknown or Not Reported | 16 | 19 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 40 | 36 | 76
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 311 | 315 | 626
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 1 | 0 | 1
Eastern Cooperative Oncology Group (ECOG) [Count of Participants; unit: Participants]
  Fully active | 261 | 267 | 528
  Restricted in physically strenuous activity | 93 | 85 | 178

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival, defined as the time from date of randomization until the earliest date of disease progression, as determined by independent central review of objective radiographic disease assessments per RECIST 1.1, or death from any cause, whichever comes first.
Time Frame: Assessed every 9 weeks for duration of study participation which is estimated to be 24 months
Population: Intent to Treat (ITT) population: consists of all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab + Epacadostat | Pembrolizumab + Placebo
Number analyzed (Participants) | 354 | 352
months | 4.7 [2.9 to 6.8] | 4.9 [2.9 to 6.8]
Statistical Analysis 1: Comparison: Pembrolizumab + Epacadostat vs Pembrolizumab + Placebo; Test type: Other; p = 0.51711, Log Rank — One-sided p-value based on log-rank test; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.83 to 1.21]

2. Primary Outcome: Overall Survival (OS) Rate at 6 Months
Description: Defined as time from date of randomization to date of death due to any cause. OS was calculated using product-limit (Kaplan-Meier) method for censored data.
Time Frame: Assessed every 9 weeks of study participation which is estimated to be 24 months. The OS rate at Month 6 was calculated.
Population: Intent to Treat (ITT) population: consists of all randomized participants. OS was analyzed at the time of primary analysis at 6 months. An overall OS was not conducted after the primary analysis since all participants were unblinded, transitioned to monotherapy pembrolizumab and survival follow-up was discontinued.
Measure: Median (95% Confidence Interval); unit: percent probability
Arm/Group | Pembrolizumab + Epacadostat | Pembrolizumab + Placebo
Number analyzed (Participants) | 354 | 352
percent probability | 84.1 [79.8 to 87.5] | 87.2 [83.2 to 90.3]
Statistical Analysis 1: Comparison: Pembrolizumab + Epacadostat; Test type: Other; p = 0.80666, Log Rank — One-sided p-value based on log-rank test; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.86 to 1.49]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response rate (ORR) is defined as the percentage of the participants in the analysis population who have a confirmed complete response (CR) or partial response (PR) based on RECIST 1.1 by independent central review.
Time Frame: Assessed every 9 weeks for duration of study participation which is estimated to be 24 months
Population: Intent to Treat (ITT) population: consists of all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Epacadostat | Pembrolizumab + Placebo
Number analyzed (Participants) | 354 | 352
Participants | 121 | 111

4. Secondary Outcome: Safety and Tolerability, as Assessed by Percentage of Participants With Adverse Events
Description: Safety and tolerability, as assessed by percentage of participants with adverse events and changes in laboratory parameters.
Time Frame: Through up to 90 days after end of treatment, up to 27 months
Population: All Subjects as Treated (ASaT): All participants who were enrolled and took at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Epacadostat | Pembrolizumab + Placebo
Number analyzed (Participants) | 353 | 352
Participants
  With one or more adverse events | 346 | 345
  Serious adverse events | 99 | 100

5. Secondary Outcome: Duration of Response (DOR)
Description: Defined as the time from the earliest date of qualifying response until earliest date of disease progression, per RECIST v1.1, or death from any cause, whichever comes first. Includes participants with complete response or partial response.
Time Frame: Assessed every 9 weeks for duration of study participation which is estimated to be 24 months
Population: Intent to Treat (ITT) population: consists of all randomized participants.
Measure: Median (Full Range); unit: months
Arm/Group | Pembrolizumab + Epacadostat | Pembrolizumab + Placebo
Number analyzed (Participants) | 354 | 352
months | NA [0.0 to NA] — Median duration not reached due to participants remaining in response at the time of the data cutoff. | NA [0.0 to NA] — Median duration not reached due to participants remaining in response at the time of the data cutoff.

6. Secondary Outcome: Apparent Oral Clearance (CL/F) of Epacadostat
Description: Defined as oral dose clearance.
Time Frame: Through up to 30 days after the end of treatment, up to 25 months
Population: All randomized participants enrolled in the Epacadostat arm currently with melanoma.
Measure: Mean (Standard Deviation); unit: Liter/hour (L/h)
Arm/Group | Pembrolizumab + Epacadostat
Number analyzed (Participants) | 340
Liter/hour (L/h) | 59.8 (17.5)

7. Secondary Outcome: Apparent Volume of Distribution (Vd/F) of Epacadostat
Description: Apparent volume of distribution after administration.
Time Frame: Through up to 30 days after the end of treatment, up to 25 months
Population: All randomized participants enrolled in the Epacadostat arm currently with melanoma.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Pembrolizumab + Epacadostat
Number analyzed (Participants) | 340
Liter | 139 (22.5)

8. Secondary Outcome: Clearance (CL) of Pembrolizumab
Time Frame: Through up to 30 days after the end of treatment, up to 25 months
Population: The data was not available nor was the analysis completed for pembrolizumab CL, because participants were unblinded and sample collections and the planned analysis for pembrolizumab CL were discontinued after the interim analysis.
Arm/Group | Pembrolizumab + Epacadostat | Pembrolizumab + Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Volume of Distribution (V) of Pembrolizumab
Time Frame: Through up to 30 days after the end of treatment, up to 25 months
Population: The data was not available nor was the analysis completed for pembrolizumab V, because participants were unblinded and sample collections and the planned analysis for pembrolizumab V were discontinued after the interim analysis.
Arm/Group | Pembrolizumab + Epacadostat | Pembrolizumab + Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Formation of Anti-pembrolizumab Antibodies
Description: Evaluate the measurement of anti-drug antibodies (ADA).
Time Frame: Through up to 30 days after the end of treatment, up to 25 months
Population: Data was not available nor the analysis completed for the incidence of ADA to pembrolizumab, because all participants were unblinded; sample collections and the planned analysis for ADA were discontinued after the interim analysis.
Arm/Group | Pembrolizumab + Epacadostat | Pembrolizumab + Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 27 months.
Description: All Subjects as Treated (ASaT): All participants who were enrolled and took at least 1 dose of study medication.
Arm/Group | Pembrolizumab + Epacadostat | Pembrolizumab + Placebo
All-Cause Mortality (participants affected / at risk) | 147/353 | 136/352
Serious Adverse Events (participants affected / at risk) | 99/353 | 100/352
Other Adverse Events (participants affected / at risk) | 327/353 | 325/352
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab + Epacadostat (N=353) | Pembrolizumab + Placebo (N=352)
Anaemia (Blood and lymphatic system disorders) | 1 | 4
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0
Extrasystoles (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 4 | 1
Hypophysitis (Endocrine disorders) | 1 | 3
Hypothyroidism (Endocrine disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Autoimmune colitis (Gastrointestinal disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 4 | 5
Diarrhoea (Gastrointestinal disorders) | 9 | 4
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Intussusception (Gastrointestinal disorders) | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 2
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 3 | 1
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 1
Death (General disorders) | 2 | 0
Fatigue (General disorders) | 1 | 2
General physical health deterioration (General disorders) | 1 | 1
Pyrexia (General disorders) | 4 | 3
Autoimmune hepatitis (Hepatobiliary disorders) | 2 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1
Dacryocanaliculitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Infected skin ulcer (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 1
Peritonitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 5 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 2
Septic shock (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0
Radiation necrosis (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 2 | 1
Blood potassium increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1
Scleroderma (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 5
Hemiplegia (Nervous system disorders) | 1 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 1
Presyncope (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 1 | 2
Tension headache (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Paranoia (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 3
Bladder outlet obstruction (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Nephritis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Renal injury (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Lichen planus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1
Essential hypertension (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 2
Lymphoedema (Vascular disorders) | 1 | 0
Retinopathy (Eye disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 | 1
Lung infection (Infections and infestations) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Carcinoid tumour of the gastrointestinal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Optic neuritis (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Bladder perforation (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab + Epacadostat (N=353) | Pembrolizumab + Placebo (N=352)
Anaemia (Blood and lymphatic system disorders) | 35 | 36
Hyperthyroidism (Endocrine disorders) | 22 | 27
Hypothyroidism (Endocrine disorders) | 44 | 35
Abdominal pain (Gastrointestinal disorders) | 37 | 37
Abdominal pain upper (Gastrointestinal disorders) | 24 | 16
Constipation (Gastrointestinal disorders) | 58 | 62
Diarrhoea (Gastrointestinal disorders) | 90 | 100
Dry mouth (Gastrointestinal disorders) | 19 | 30
Nausea (Gastrointestinal disorders) | 103 | 86
Vomiting (Gastrointestinal disorders) | 51 | 44
Asthenia (General disorders) | 68 | 46
Fatigue (General disorders) | 100 | 94
Oedema peripheral (General disorders) | 27 | 27
Pyrexia (General disorders) | 46 | 38
Nasopharyngitis (Infections and infestations) | 50 | 50
Upper respiratory tract infection (Infections and infestations) | 19 | 33
Urinary tract infection (Infections and infestations) | 20 | 32
Alanine aminotransferase increased (Investigations) | 39 | 25
Amylase increased (Investigations) | 27 | 34
Aspartate aminotransferase increased (Investigations) | 36 | 33
Lipase increased (Investigations) | 36 | 39
Weight decreased (Investigations) | 22 | 17
Decreased appetite (Metabolism and nutrition disorders) | 55 | 44
Hyperglycaemia (Metabolism and nutrition disorders) | 23 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 63 | 63
Back pain (Musculoskeletal and connective tissue disorders) | 47 | 52
Myalgia (Musculoskeletal and connective tissue disorders) | 26 | 32
Pain in extremity (Musculoskeletal and connective tissue disorders) | 32 | 28
Dizziness (Nervous system disorders) | 33 | 32
Headache (Nervous system disorders) | 66 | 74
Anxiety (Psychiatric disorders) | 19 | 14
Insomnia (Psychiatric disorders) | 35 | 31
Cough (Respiratory, thoracic and mediastinal disorders) | 73 | 63
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 | 29
Dry skin (Skin and subcutaneous tissue disorders) | 23 | 23
Pruritus (Skin and subcutaneous tissue disorders) | 83 | 101
Rash (Skin and subcutaneous tissue disorders) | 77 | 81
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 21 | 18
Vitiligo (Skin and subcutaneous tissue disorders) | 51 | 48
Hypertension (Vascular disorders) | 27 | 21
Influenza (Infections and infestations) | 19 | 17
Influenza like Illness (General disorders) | 17 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-18): https://cdn.clinicaltrials.gov/large-docs/74/NCT02752074/Prot_SAP_000.pdf